CLINICAL TRIAL: NCT06634459
Title: The POMEGRANATE Trial: A Randomized Controlled Trial Comparing Pessary Home Management of Reia Pessary Versus Standard of Care Pessary for Treatment of Pelvic Organ Prolapse
Brief Title: POMEGRANATE Trial: Comparing Reia Pessary Versus Standard of Care Pessary for Pelvic Organ Prolapse Treatment
Acronym: POMEGRANATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POM-110
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Organ Prolapse; Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either (1) the Reia System (RS) or (2) standard pessary care (SPC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reia System (Active Comparator): Participants receiving the commercially available RS will be fit with one of three available pessary sizes and will receive an applicator corresponding to their pessary size.
  Interventions: Device: Reia System
- Standard Pessary Care (Active Comparator): Participants receiving SPC will be fit with a Gellhorn pessary or ring with/without support without knob pessary per standard clinical protocol.
  Interventions: Device: Standard of Care Pessary

INTERVENTIONS:
Device: Reia System — Reia pessary
  Arms: Reia System
Device: Standard of Care Pessary — Gellhorn pessary or ring with/without support without knob pessary
  Arms: Standard Pessary Care

SUMMARY:
This multi-centered, randomized controlled trial will evaluate the safety and efficacy of home use of the novel Reia System (RS), which includes the Reia pessary and applicator, compared to standard pessary care (Gellhorn or ring with/without support without knob) among women with stage II-IV pelvic organ prolapse (POP). A total of 182 participants will be recruited among pessary naïve patients who are symptomatic and choose a vaginal pessary for management of their POP from study sites specializing in Urogynecology and Reconstructive Pelvic Surgery (URPS). Participants will be assigned via 1:1 randomization using computer generated numbers in permutated groups of variable block sizes to either the intervention (the Reia System, RS) or standard pessary care (SPC) stratified by site. Participation in this trial will involve a total of four visits over six months. The primary outcome measure will be satisfaction measured at the six-month time point. Secondary outcomes will include validated surveys to assess quality of life, number of self-management events, ease/difficulty of pessary insertion/removal, importance of ability to self-manage pessary, and adverse events.

Specific Aims

Aim 1: To compare satisfaction with pessary use and management between subjects randomized to the Reia System and those randomized to standard of care pessary.

Aim 2: To assess successful fitting, number of refitting visits, number of self-management events and continued pessary use over a 6-month period between subjects randomized to the Reia System and those randomized to standard of care pessary.

Aim 3: To compare ease/difficulty of pessary use and importance of ability to self-manage, as well as quality of life over a 6-month period between subjects randomized to the Reia System and those randomized to standard of care pessary.

Aim 4: To measure rates of adverse events and risk factors for adverse events over a 6-month period between subjects randomized to the Reia System and those randomized to standard of care pessary.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking natal females ≥ 18 years of age
* Willing to self-maintain (insert/remove) pessary
* Pessary naïve with Stage II-IV POP desiring conservative management with a pessary
* Primary indication for use of pessary is treatment of pelvic organ prolapse

Exclusion Criteria:

* Primary indication for pessary use is for management of stress urinary incontinence
* Prior mesh-augmented prolapse repair (i.e. transvaginal mesh, sacrocolpopexy)
* Short vaginal length (TVL < 8cm) or subjective vaginal narrowing
* Vaginal fistula (e.g. rectovaginal, vesicovaginal or any type of fistula involving the vagina)
* Vaginal, rectal or bladder malignancy
* Genitourinary infection requiring treatment (See below 1)
* Ongoing treatment for vaginal infections (e.g., chronic bacterial vaginosis) (See below 2)
* Inflammatory bowel disease (Crohn's or ulcerative colitis)
* Pelvic or anorectal chronic pain
* Pelvic floor surgery within the past 6 months or planning to undergo pelvic floor surgery
* Congenital malformation of the bladder, rectum or vagina
* Pregnant or planning pregnancy in the next 6 months
* Prior failure of pessary for POP
* History of hydroureter, hydronephrosis, or impaired renal function secondary to prolapse

  1. Patients with acute vaginal infections will be eligible for enrollment 2 weeks after completing treatment with resolution of symptoms
  2. OK to be on prophylactic/suppressive therapy for HSV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with treatment | 6 months
  The primary outcome will be measured by participant response to the question "How satisfied or unsatisfied are you with your ability to use and manage the pessary provided to you?" with response collected via VAS ranging from "0mm = very unsatisfied" to "100mm = very satisfied" with 50mm = neutral (neither satisfied nor unsatisfied).

SECONDARY OUTCOMES:
Total self-management events | 6 months
  Defined as removing the pessary ≥ one time per 24-hour period over the six-month follow-up period, this outcome will be summed and divided by actual days of follow-up to accommodate minor variation across participants in the exact length of follow-up.
Patient Global Impression of Severity (PGI-S) | 6 months
  A single item questionnaire to assess the patient's impression of disease severity. For purposes of this trial, the investigators have adapted the PGI-I to specifically ask about "prolapse" severity. It will ask participants to "Check the one number that best describes how the participant's prolapse condition is now" on a 4-point Likert scale ranging from (1) normal to (4) severe
Patient Global Impression of Improvement (PGI-I) | 6 months
  A single item questionnaire to assess a patient's impression of change. For purposes of this trial, the investigators have adapted the PGI-I to specifically ask about "prolapse symptoms." It will ask participants to "Check the one number that best describes how the participant's prolapse condition is now, compared with how it was before the participant began this study" on a 7-point Likert scale ranging from (1) very much better to (7) very much worse
Pelvic Floor Distress Inventory-20 (PFDI-20) | 6 months
  A 20-item condition-specific quality-of-life instrument with three scales (6-item Urinary Distress Inventory, 6-item Pelvic Organ Prolapse Distress Inventory, and 8-item Colorectal-Anal Distress Inventory) used to evaluate the impact of pelvic floor disorders on quality of life with a response scale from 0 (not present) to 4 (quite a bit bothersome).
Pelvic Floor Impact Questionnaire-7 (PFIQ-7) | 6 months
  A 7-item condition-specific quality-of-life instrument with three scales (Urinary, Pelvic Organ Prolapse, and Colorectal-Anal). The PFIQ-7 is a validated instrument that is widely utilized in research in conjunction with the PFDI-20 to provide a comprehensive evaluation of the impact of pelvic floor disorders on quality of life, specifically how they affect activities, relationships, and feelings on a scale from not at all to quite a bit.
Patient Global Symptoms Control Rating Scale (PGSC) | 6 months
  A a single item adapted for purposes of this trial. It will state "My current treatment is giving me adequate control of my prolapse" and participants will be asked to select a response on a 5-point Likert scale ranging from (1) disagree strongly to (5) agree strongly
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) | 6 months
  A validated instrument to evaluate sexual function in women with pelvic organ prolapse and/or urinary incontinence with 21 questions for sexually active women and 12 questions for non-sexually active women
Pessary outcomes | 6 months
  Will include continued use of pessary and number of unintentional pessary expulsions
Behavioral Outcomes | 6 months
  Will include a 5-point Likert scale ranging from (1) disagree strongly to (5) agree strongly about participants' ease of self-administered pessary insertion, ease of self-administered pessary removal, discomfort with self-administration of pessary insertion, and discomfort with self-administration of pessary removal
Participant view of importance of ability to self-maintain pessary | 6 months
  This outcome will be measured by the question "How important is it to you to be able to self-manage your pessary?" with response options on a 5-point Likert scale of 1-not at all important, 2-slightly important, 3-neutral, 4-moderately important, 5-very important.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - MedStar Health, Washington D.C., District of Columbia
  - The University of Chicago, Northbrook, Illinois
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Women & Infants Hospital in Rhode Island, Providence, Rhode Island
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Constantine ML, Pauls RN, Rogers RR, Rockwood TH. Validation of a single summary score for the Prolapse/Incontinence Sexual Questionnaire-IUGA revised (PISQ-IR). Int Urogynecol J. 2017 Dec;28(12):1901-1907. doi: 10.1007/s00192-017-3373-9. Epub 2017 Jun 6. PMID 28589290
- [Background] Rogers RG, Rockwood TH, Constantine ML, Thakar R, Kammerer-Doak DN, Pauls RN, Parekh M, Ridgeway B, Jha S, Pitkin J, Reid F, Sutherland SE, Lukacz ES, Domoney C, Sand P, Davila GW, Espuna Pons ME. A new measure of sexual function in women with pelvic floor disorders (PFD): the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1091-103. doi: 10.1007/s00192-012-2020-8. Epub 2013 Apr 30. PMID 23632798
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] R Core. R Core Team (2020). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. Accessed December 20, 2021.
- [Background] Pinhero J, Bates D. Mixed Effects Models in S and S-plus: Springer; 2000.
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Background] Health UDo, Services H. Common Terminology Criteria for Adverse Events. Version 5.0. Published November 27, 2017. 2020.
- [Background] Strohbehn K, Wadensweiler P, Hanissian P. A novel, collapsible, space-occupying pessary for the treatment of pelvic organ prolapse. Int Urogynecol J. 2023 Jan;34(1):317-319. doi: 10.1007/s00192-022-05415-y. Epub 2022 Dec 3. No abstract available. PMID 36462059
- See also: Related Info — https://www.r-project.org.